CLINICAL TRIAL: NCT02723604
Title: A Phase II Prospective Trial of Low-Level Laser Therapy for Prevention of Oral Mucositis in Patients Receiving Chemotherapy and Radiation for Head and Neck Cancer
Brief Title: Low-Level Laser Therapy for Prevention of Oral Mucositis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Harold Kim, Principal Investigator, Barbara Ann Karmanos Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2015-170; NCI-2016-00406 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2015-170 (Other: Wayne State University/Karmanos Cancer Institute); P30CA022453 (NIH)
Record Dates: First submitted 2016-03-21; First posted 2016-03-30 (Estimated); Results first posted 2023-02-27 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: Mucositis
MeSH Terms: conditions — Mucositis | interventions — Low-Level Light Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Experimental: Low Level Laser Therapy (Experimental): Patients meeting the eligibility criteria will be enrolled to receive prophylactic LLLT in addition to standard of care measures for oral mucositis or other toxicity of therapy. The radiation and chemotherapy dose, schedule, modality, technique, and any required adjustments will not be influenced by this protocol and will follow standard existing institutional practices.
  Interventions: Device: Low Level Laser Therapy

INTERVENTIONS:
Device: Low Level Laser Therapy — Patients will receive LLLT three times per week concurrently with chemoradiotherapy. LLLT may be delivered either immediately prior to or after the patient's daily fraction of radiotherapy. Patients will be treated extra-orally with a THOR® LED cluster for one minute along the buccal mucosa on each side and intraorally for one minute to the tongue and soft palate. During each LLLT treatment session a thorough oral exam will be performed to identify any areas of mucositis. If the patient should develop intraoral lesions they will be targeted directly with the intraoral probe for one minute to each site of mucositis. The laser settings to be used are as follows: frequency 2.5 Hz; wavelength 660 nm; and power 75 mW, for an energy of 4.5 J.

SUMMARY:
The overall purpose of this study is to examine the efficacy of prophylactic low-level laser therapy (LLLT) to reduce the incidence of oral mucositis and adverse events in patients receiving combined modality therapy consisting of chemotherapy and radiation therapy for head and neck cancer.

DETAILED DESCRIPTION:
A phase II, single-arm trial to examine the efficacy of prophylactic low-level laser therapy (LLLT) to reduce the incidence of oral mucositis and adverse events in patients receiving combined modality therapy consisting of chemotherapy and radiation therapy for head and neck cancer.

Patients meeting the eligibility criteria will be enrolled to receive prophylactic LLLT in addition to standard of care measures for oral mucositis or other toxicity of therapy. The radiation and chemotherapy dose, schedule, modality, technique, and any required adjustments will not be influenced by this protocol and will follow standard existing institutional practices.

Patients will receive LLLT three times per week concurrently with chemoradiotherapy. LLLT may be delivered either immediately prior to or after the patient's daily fraction of radiotherapy. Patients will be treated extra-orally with a THOR® LED cluster for one minute along the buccal mucosa on each side and intraorally for one minute to the tongue and soft palate. During each LLLT treatment session a thorough oral exam will be performed to identify any areas of mucositis. If the patient should develop intraoral lesions they will be targeted directly with the intraoral probe for one minute to each site of mucositis. The laser settings to be used are as follows: frequency 2.5 Hz; wavelength 660 nm; and power 75 mW, for an energy of 4.5 J.

Patients will be evaluated prior to therapy, weekly during therapy, two weeks after the completion of therapy, and three months after the completion of therapy. During each assessment, the following toxicities will be assessed: pain, mucositis, dysphagia, xerostomia, dysgeusia, dermatitis, trismus, and quality of life.

Previous studies indicate that approximately 40% of patients will experience severe mucositis with radiation and concurrent chemotherapy. The hypothesis in this trial is that the addition of LLLT to this treatment regimen will decrease the rate of severe acute oral mucositis (OM) to 20%. We plan to enroll 25 patients at our institution in 12 months after the trial opens.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to understand and sign informed consent form approved by the institutional review board (IRB)
* Males or females greater than or equal to 18 years old
* Biopsy-proven head and neck cancer (HNC) including cancers of the nasopharynx, oropharynx, larynx, hypopharynx, or HNC of unknown primary origin amenable to therapy with radiation and concurrent chemotherapy
* Patients who are planned to receive definitive or adjuvant radiotherapy with concurrent platinum-based chemotherapy
* Patients whose clinical treatment plans include a continuous course of external beam radiotherapy by intensity-modulated radiation therapy (IMRT) and/or image-guided radiation therapy (IGRT), given as a cumulative dose of 5000 - 7000 centigray (cGy) in single daily fractions of 180 - 200 cGy, combined with a concurrent course of weekly or tri-weekly cisplatin or carboplatin chemotherapy
* Karnofsky performance status score > 60
* Female patients of child-bearing potential must have a negative pregnancy test prior to enrollment

Exclusion Criteria:

* Patient has evidence of current mucositis, mucosal ulceration, or unhealed surgical wounds from surgical resection or biopsy
* Prior radiation to the head and neck
* Patients with gross tumor involvement of the oral cavity or oral mucosa
* Patient planned to receive altered fractionation radiotherapy or multiple fractions per day
* Patient is using a pre-existing feeding tube for nutritional support at the time of study entry
* Women who are pregnant or breast-feeding
* Patient plans to receive concurrent chemotherapy, other than the regimens specified in the inclusion criteria
* Patients who have chronic immunosuppression or are on current immunosuppressive therapies
* Patients who have a contraindication to radiation therapy
* Patients enrolled on another investigational trial for oral mucositis prevention
* Life expectancy of less than 3 months
* Unable or unwilling to adhere to study-specified procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2016-03; Primary Completion 2017-08-02 (Actual); Study Completion 2021-09-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harold Kim, Principal Investigator — Barbara Ann Karmanos Cancer Institute
Locations (1):
- Wayne State University/Karmanos Cancer Institute, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
The same protocol will be opened separately at the University of Pittsburgh Medical Center, where an additional 25 patients will be enrolled. A Data Use Agreement will allow combination of the data for a total of 50 patients to be analyzed.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Experimental: Low Level Laser Therapy
Started | 25
Completed | 23
Not Completed | 2
Not completed — ineligible | 1
Not completed — never received treatment | 1

BASELINE CHARACTERISTICS:
Arm/Group | Experimental: Low Level Laser Therapy
Number analyzed (Participants) | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.5 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 18
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 23

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Severe (Common Terminology Criteria for Adverse Events Version 4.0 [CTCAE v. 4.0] Grade 3-5 Oral Mucositis in Patients Treated to a Cumulative Radiation Dose of at Least 5000 cGy
Time Frame: From beginning of therapy up to 3 months after completion of therapy
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental: Low Level Laser Therapy
Number analyzed (Participants) | 23
Participants | 15

2. Primary Outcome: Number of Participants With Severe World Health Organization [WHO] (Grade 3-4) Oral Mucositis in Patients Treated to a Cumulative Radiation Dose of at Least 5000 cGy
Time Frame: From beginning of therapy up to 3 months after completion of therapy
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental: Low Level Laser Therapy
Number analyzed (Participants) | 23
Participants | 10

3. Secondary Outcome: Change in OM-related QOL Assessed Using FACT Questionnaire
Description: The QOL assessment taken at the beginning of therapy is subtracted from the QOL assessment taken at the completion of therapy. The QOL scale is the FACT Questionnaire. Measure on a scale of 0 to 4. 0 = not at all and 4= very much.
Time Frame: From beginning of therapy up to completion of therapy
Population: 5 patients were missing either the beginning and/or completion of therapy QOL data
Measure: Mean (90% Confidence Interval); unit: units on a scale
Arm/Group | Experimental: Low Level Laser Therapy
Number analyzed (Participants) | 18
units on a scale | 2.3 [1.9 to 2.8]

4. Secondary Outcome: Duration of Oral Mucositis
Description: Survival analysis was used to estimate the duration of oral mucositis. Patients were censored if oral mucositis not resolved by the end of the study.
Time Frame: From beginning of therapy up to 3 months after completion of therapy
Population: 15 of the 23 patients had at least 1 episode of oral mucositis. 2 patients had 2 distinct episodes of oral mucositis. Each instance was analyzed separately
Measure: Median (90% Confidence Interval); unit: weeks
Units Other Than Participants: instances
Arm/Group | Experimental: Low Level Laser Therapy
Number analyzed (Participants) | 15
Number analyzed (instances) | 17
weeks | 4 [4 to NA] — Kaplan-Meier estimation was used for this analysis. The 90% upper limit of the confidence interval did not cross 50%.

5. Secondary Outcome: Number of Participants With Any Grade Oral Mucositis in Patients Treated to a Cumulative Radiation Dose of at Least 5000 cGy
Description: Grade of oral mucositis assessed using the NCI CTCAE version 4.0
Time Frame: From beginning of therapy up to 3 months after completion of therapy
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental: Low Level Laser Therapy
Number analyzed (Participants) | 23
Participants | 23

6. Secondary Outcome: Number of Participants With Dysgeusia Assessed by CTCAE v. 4.0
Description: Variable is reported on the 1-5 CTCAE scale:
  1. - Mild
  2. - Moderate
  3. - Severe
  4. - Life-threatening
  5. - Death
  The maximum recorded severity is reported.
Time Frame: From beginning of therapy up to 3 months after completion of therapy
Measure: Number; unit: participants
Arm/Group | Experimental: Low Level Laser Therapy
Number analyzed (Participants) | 23
participants
  Grade 1 | 0
  Grade 2 | 23
  Grade 3 | 0
  Grade 4 | 0
  Grade 5 | 0

7. Secondary Outcome: Number of Participants With Dysphagia Assessed by CTCAE v. 4.0 and Diet Assessment
Description: as for outcome 6
Time Frame: From beginning of therapy up to 3 months after completion of therapy
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental: Low Level Laser Therapy
Number analyzed (Participants) | 23
Participants
  Grade 1 | 2
  Grade 2 | 17
  Grade 3 | 4
  Grade 4 | 0
  Grade 5 | 0

8. Secondary Outcome: Number of Participants With Pain as Assessed by the Visual Analogue Scale (VAS)
Description: Variable is reported on the 1-10 scale Higher values represent a worse outcome The maximum recorded severity is reported
Time Frame: From beginning of therapy up to 3 months after completion of therapy
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental: Low Level Laser Therapy
Number analyzed (Participants) | 23
Participants
  1 | 0
  2 | 0
  3 | 2
  4 | 0
  5 | 5
  6 | 2
  7 | 2
  8 | 5
  9 | 4
  10 | 3

9. Secondary Outcome: Number of Participants With Radiodermatitis Assessed by CTCAE v. 4.0
Description: as for outcome 6
Time Frame: From beginning of therapy up to 3 months after completion of therapy
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental: Low Level Laser Therapy
Number analyzed (Participants) | 23
Participants
  Grade 1 | 5
  Grade 2 | 16
  Grade 3 | 2
  Grade 4 | 0
  Grade 5 | 0

10. Secondary Outcome: Number of Participants With Trismus Assessed by Measurement of Interincisal Distance
Description: Trismus is defined as a measurement of interincisal distance less than or equal to 30mm.
Time Frame: From beginning of therapy up to 3 months after completion of therapy
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental: Low Level Laser Therapy
Number analyzed (Participants) | 23
Participants | 2

11. Secondary Outcome: Number of Participants With Xerostomia Assessed by CTCAE v. 4.0
Description: as for outcome 6
Time Frame: Up to 3 months after completion of therapy
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental: Low Level Laser Therapy
Number analyzed (Participants) | 23
Participants
  Grade 1 | 2
  Grade 2 | 17
  Grade 3 | 4
  Grade 4 | 0
  Grade 5 | 0

12. Secondary Outcome: Mean Cumulative Radiation Dose at Time of Onset of Severe (CTCAE v. 4.0 Grade 3-4) Oral Mucositis
Description: The reported dose is at the first incidence of severe oral mucositis.
Time Frame: From beginning of therapy up to 3 months after completion of therapy
Population: 15 patients had severe oral mucositis; 3 were missing dose information
Measure: Mean (90% Confidence Interval); unit: Gray
Arm/Group | Experimental: Low Level Laser Therapy
Number analyzed (Participants) | 12
Gray | 53.5 [47.68 to 59.32]

13. Secondary Outcome: Time to Onset of Severe (CTCAE v. 4.0 Grade 3-4) Oral Mucositis Following the Initiation of Radiotherapy
Description: Survival analysis is used to analyze this endpoint
Time Frame: From beginning of therapy up to 3 months after completion of therapy
Measure: Median (90% Confidence Interval); unit: weeks
Arm/Group | Experimental: Low Level Laser Therapy
Number analyzed (Participants) | 23
weeks | NA [7 to NA] — The Kaplan-Meier curve and upper confidence limit did not cross 50%

14. Other Pre Specified Outcome: Amount of Narcotic Analgesia Use During Treatment
Time Frame: From beginning of therapy up to 3 months after completion of therapy
Population: Data not collected
Arm/Group | Experimental: Low Level Laser Therapy
Number analyzed (Participants) | 0

15. Other Pre Specified Outcome: Number of Participants With Breaks in Treatment
Description: Breaks in treatment defined as one of the following: Missing at least 1 chemotherapy treatment; dose reduction in planned cisplatin administration; OR 3 consecutive days of no radiation therapy secondary to mucositis
Time Frame: Date of completion of chemoradiation therapy
Population: Data not collected
Arm/Group | Experimental: Low Level Laser Therapy
Number analyzed (Participants) | 0

16. Other Pre Specified Outcome: Percent Change in Body Weight During the Course of Treatment
Description: The percent change in body weight was computed by subtracting the baseline weight from the weight after completion of treatment and dividing that quantity by the baseline weight. The confidence interval is estimated using the t distribution.
Time Frame: From date of enrollment until the date of completion of chemoradiation therapy, assessed up to 3 months after completion of therapy
Measure: Number (90% Confidence Interval); unit: percent change in body weight
Arm/Group | Experimental: Low Level Laser Therapy
Number analyzed (Participants) | 23
percent change in body weight | -10.9 [-13.0 to -8.7]

17. Other Pre Specified Outcome: Number of Participants Who Require Feeding Tube Placement During Treatment (Excluding Patients Who Received a Prophylactic Feeding Tube Prior to the Initiation of Therapy)
Time Frame: At the date of completion of chemoradiation therapy
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental: Low Level Laser Therapy
Number analyzed (Participants) | 23
Participants | 7

18. Other Pre Specified Outcome: Number of Participants With Severe (CTCAE v. 4.0 Grade 3-4) Oral Mucositis by 5000 and 7000 cGy
Time Frame: From beginning of therapy up to 3 months after completion of therapy
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental: Low Level Laser Therapy
Number analyzed (Participants) | 23
Participants
  Treated with 70Gy & had OM | 14
  Treated with 70Gy & did not have OM | 6
  Treated with 50-69Gy & had OM | 1
  Treated with 50-69Gy & did not have OM | 2

19. Other Pre Specified Outcome: Number of Participants With Severe (CTCAE v. 4.0 Grade 3-4) Oral Mucositis by Schedule of Chemotherapy Given Weekly Versus Every 3 Weeks
Time Frame: From beginning of therapy up to 3 months after completion of therapy
Population: Data not collected
Arm/Group | Experimental: Low Level Laser Therapy
Number analyzed (Participants) | 0

20. Other Pre Specified Outcome: Time to Reach Planned Dose of Radiation Therapy
Description: Kaplan-Meier methods are used to estimate time until reaching planned dose.
Time Frame: From the beginning of therapy up to completion of therapy (9 weeks maximum)
Population: 1 patient is missing dose information; 5 did not reach planned dose
Measure: Median (Full Range); unit: weeks
Arm/Group | Experimental: Low Level Laser Therapy
Number analyzed (Participants) | 17
weeks | 9 [8 to 9]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from the beginning of treatment, up until 3 months after the completion of treatment.
Arm/Group | Experimental: Low Level Laser Therapy
All-Cause Mortality (participants affected / at risk) | 0/23
Serious Adverse Events (participants affected / at risk) | 0/23
Other Adverse Events (participants affected / at risk) | 23/23
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental: Low Level Laser Therapy (N=23)
Dysphagia (General disorders) | 23 (23)
Xerostomia (General disorders) | 23 (23)
Dysgeusia (General disorders) | 23 (23)
Trismus (General disorders) | 2 (2)
Radiodermatitis (General disorders) | 23 (23)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-07-20): https://cdn.clinicaltrials.gov/large-docs/04/NCT02723604/Prot_SAP_000.pdf